CLINICAL TRIAL: NCT00978705
Title: Clinical Study for Evaluation of Clinical Efficacy and Safety of Autologous Cultured Keratinocyte Cell on Severe Burn Wood
Brief Title: Clinical Efficacy and Safety of Autologous Cultured Keratinocyte Cell on Severe Burn Wood
Acronym: keratinocyte
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Biosolution Co., Ltd. (Industry)
Responsible Party: Yunyoung Kim / Senior Research Scientist, Modern Cell and Tissue Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCTT-KRH-06
Record Dates: First submitted 2009-04-15; First posted 2009-09-17 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Burn Wound
Keywords: Keratinocyte Cell; severe burn wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Autologous cultured keratinocyte cell — 3x10^7 cell/ vial
  Other Names: Keraheal

SUMMARY:
The efficacy and safety of Autologous cultured keratinocyte cell on severe burn wound.

ELIGIBILITY:
Inclusion Criteria:

* Age : 1~70 years
* More than 30% TBSA of second degree burn or more than 10% TBSA of third degree burn
* Must provide signed informed consent prior to participation in any study-related procedures

Exclusion Criteria:

* Have a pyogenic infection
* Part of the facial cosmetic surgery cost
* Hypersensitivity reactions in patients with bovine proteins
* Hypersensitivity reactions in patients with Gentamycin
* Pregnancy or lactation

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-05 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
engraftment assessment | 4week

SECONDARY OUTCOMES:
the vancouver burn scar scale | 8, 12, 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Wook Chun, MD, Principal Investigator — Hangang Sacred Heart Hospital
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, South Korea